CLINICAL TRIAL: NCT02182739
Title: Programa de Experiencia Therapéutica Personalizada (Personalized Therapeutic Experience Program)
Brief Title: Observational Study of Meloxicam in Any Labeled Indication
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 107.249
Record Dates: First submitted 2014-07-03; First posted 2014-07-08 (Estimated); Last update posted 2014-10-29 (Estimated); Status verified 2014-07

CONDITIONS: Arthritis, Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Meloxicam

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Meloxicam
  Interventions: Drug: Meloxicam

INTERVENTIONS:
Drug: Meloxicam — tablets or injectable solution

SUMMARY:
Evaluation on the amelioration of symptom intensity of the indication and to evaluate drug tolerability.

ELIGIBILITY:
Inclusion Criteria:

* Patients according to the physicians medical criteria on the labeled indications for Meloxicam

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: primary care
Sampling Method: Non-Probability Sample
Enrollment: 13039 (Actual)
Dates: Start 2001-01; Primary Completion 2001-12 (Actual)

PRIMARY OUTCOMES:
Change in assessment of intensity of pain on a 4-point verbal rating scale | up to 1 year
Assessment of tolerability on a 4-point scale | up to 1 year

SECONDARY OUTCOMES:
Number of patients with adverse events | up to 1 year